CLINICAL TRIAL: NCT00177580
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial of Adjunctive Treatment With Pravastatin in Partially Remitted Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Improving Symptoms of Schizophrenia and Schizoaffective Disorder by Supplementing Medications With Pravastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0308022
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; positive symptoms; negative symptoms; cognitive functioning; pravastatin
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pravastatin

INTERVENTIONS:
Drug: Pravastatin

SUMMARY:
This study supplements patients' current medications with Pravastatin, a cholesterol-lowering medication, to try to improve residual symptoms of schizophrenia, and also to improve cognitive functioning.

DETAILED DESCRIPTION:
This study supplements patients' current medications with Pravastatin, a cholesterol-lowering medication, to try to improve residual symptoms and also to improve cognitive functioning. It consists of 15 total study visits over a 28-week period of time, one visit every 2 weeks.

Blood draws will be done once every 4 weeks throughout the study to monitor lipid levels, C-Reactive protein, AST, ALT, and CPK Total. Cognitive testing will be completed at the beginning of the study and at the end of the study. During the study visits, the staff will be monitoring vitals signs (weight, height, blood pressure, pulse, waist/hip ratio), possible side effects, positive and negative symptoms, mood symptoms, and overall functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Male and female subjects; age 18-65 years inclusive
* Ability to provide informed consent
* No psychiatric hospitalization in the last 30 days prior to randomization
* PANSS score at study entry between 80 and 120 inclusive, OR those who continue to experience some residual positive and/or negative symptoms and are not at their baseline level of functioning.
* Current psychiatric medications stable for at least 30 days
* Currently receiving only one antipsychotic medication
* Female subjects of child-bearing age must use an acceptable method of birth control

Exclusion Criteria:

* Active, uncontrolled, or chronic liver disease
* Heart failure
* Current alcohol abuse or dependence
* Female subjects who are pregnant, lactating or plan to become pregnant during the study period
* History of allergic reaction with any statin in the past
* Kidney disorder or other evidence of renal dysfunction
* Uncontrolled diabetes
* Untreated hyperlipidemia
* Concurrently receiving treatment with cyclosporine, gemfibrozil, clofibrate, fenofibrate, niacin, macrolide antibiotics, erythromycin, HIV protease inhibitors, nefazodone, or verapamil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
PANSS total score (clinical state)

SECONDARY OUTCOMES:
Safety
Positive Symptoms
Negative Symptoms
Depressive Symptoms
Cognitive Functions
Social Functioning
C-Reactive Protein changes
Lipid Enzyme changes

CONTACTS AND LOCATIONS:
Overall Officials: Jaspreet S Brar, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: This website describes the pravastatin research study, and describes the purpose of our research program. — http://www.wpic.pitt.edu/research/SWRP/